CLINICAL TRIAL: NCT02913911
Title: The Provision of External Feedback During Sit-to-stand in Ambulatory Patients With Spinal Cord Injury
Brief Title: Sit-to-stand With Feedback in SCI Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Sugalya Amatachaya, Assoc. Prof. Dr., Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2559A10303150
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2015-11

CONDITIONS: Injuries, Spinal Cord
Keywords: feedback
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback (Experimental): Subjects will be trained using the sit-to-stand weight-taking machine. Prior to the training, subjects sit in a standard sitting position. Then they will be instructed to take most of their body-weight onto the legs while they standing up where the light bars will be gradually lightened from the red, yellow and green zones according to the level of LLL. Then they stand up, hold a standing position for 3-5 seconds and sit-down with always maximize their body-weight onto their legs during performing the task in which the green zone will always be lightened.
  Interventions: Other: feedback
- No feedback (Sham Comparator): Subjects will be trained using the same instruction and protocol as the experimental group, but without the provision of external feedback.
  Interventions: Other: feedback

INTERVENTIONS:
Other: feedback — Sit to stand training with external feedback

SUMMARY:
* Does the utility of external feedback in terms of goal-directed LLL approach during STS training immediately improve functional ability relating to walking in ambulatory patients with SCI?
* Does the utility of LLL feedback improve functional ability relating to walking in ambulatory patients with SCI after 2-week training?

DETAILED DESCRIPTION:
* To compare immediate effects of STS training with and without LLL feedback on functional ability relating to walking in ambulatory patients with SCI
* To compare 2 weeks effects of STS training with and without LLL feedback on functional ability relating to walking in ambulatory patients with SCI.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory spinal cord injury patients

Exclusion Criteria:

* Deformity of musculoskeletal system

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
10MWT | 2 weeks
  walking speed test

CONTACTS AND LOCATIONS:
Overall Officials: Sugalya Amatachaya, Ph.D., Principal Investigator — School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No